CLINICAL TRIAL: NCT00254969
Title: Immunogenicity and Safety of Pentaxim in South African Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E2I43
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Diphtheria; Tetanus; Haemophilus Infections; Pertussis; Poliomyelitis
Keywords: Diphteria; tetanus; haemophilus influenzae type b; poliomyelitis; pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Haemophilus Infections; Whooping Cough; Poliomyelitis | interventions — Tetanus Toxoid; Pentavac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Diphtheria, Tetanus, Polio, Acellular Pertussis and Hib

INTERVENTIONS:
Biological: Diphtheria, Tetanus, Polio, Acellular Pertussis and Hib — 0.5 mL, Im
  Other Names: PENTAXIM™

SUMMARY:
The present clinical study will assess the immunogenicity and reactogenicity of Aventis Pasteur's DTacP-IPV// PRP~T combined vaccine (Pentavac™ or Pentaxim™) as a three-dose primary vaccination at 6, 10 and 14 weeks of age followed by a booster dose during the second year of life in order to meet the requirements for application for the use of the product in the Expanded Program on Immunization (EPI) in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Aged < 24 hours on the day of inclusion

Exclusion Criteria:

* At visit 01 (screening)
* Illness at a stage that could interfere with trial conduct or completion.
* Any vaccination preceding the trial participation (except Bacille Calmette-Guerin [BCG])
* Acute illness on the day of screening. At visit 01 and visit 02 (screening and first study vaccination).
* Planned participation in another clinical trial during the present trial period
* Blood or blood-derived products received since birth.
* Mother known as seropositive to HIV or hepatitis B.
* Known thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of/current seizures at visit 02 (first study vaccination)
* Participation in another clinical trial preceding the first trial vaccination
* Congenital or acquired immunodeficiency; immunosuppressive therapy such as long-term systemic corticosteroid therapy.
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Any vaccination preceding the first trial vaccination (except BCG)
* History of diphtheria, tetanus, pertussis, poliomyelitis, Haemophilus influenzae type b and hepatitis B infection (confirmed either clinically, serologically or microbiologically).
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, Haemophilus influenzae type b and hepatitis B infection with the trial vaccine or another vaccine.
* Febrile illness (rectal temperature ≥ 38.0°C or axillary temperature ≥ 37.4°C) or acute illness on the day of first vaccination

Min Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of DTacP-IPV//PRP~T combined vaccine. | 1 month post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Soweto, South Africa

REFERENCES:
- [Derived] Madhi SA, Cutland C, Jones S, Groome M, Ortiz E. One-year post-primary antibody persistence and booster immune response to a DTaP-IPV//PRP~T vaccine (Pentaxim) given at 18 - 19 months of age in South African children primed at 6, 10 and 14 weeks of age with the same vaccine. S Afr Med J. 2011 Nov 28;101(12):879-83. PMID 22273029
- See also: Related Info — http://www.sanofipasteur.com